CLINICAL TRIAL: NCT03764527
Title: Randomized Study of the Tolerability and Efficacy of Artemether-Lumefantrine Versus Artesunate Plus Amodiaquine Coadministered for the Treatment of Uncomplicated Falciparum Malaria in Zanzibar
Brief Title: Tolerability and Efficacy of Artemether-Lumefantrine Versus Artesunate + Amodiaquine in Zanzibar
Acronym: AcoI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Professor Anders Björkman (Other)
Collaborators: Zanzibar Malaria Control Programme (Other Government); World Health Organization (Other)
Responsible Party: Sponsor-Investigator, Professor Anders Björkman, Professor, Karolinska Institutet
Organization: Karolinska Institutet (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Aco-study
Record Dates: First submitted 2018-12-03; First posted 2018-12-05 (Actual); Last update posted 2018-12-06 (Actual); Status verified 2018-12

CONDITIONS: Plasmodium Falciparum Malaria
Keywords: Artemether-Lumefantrine; Coartem; Artesunate; Amodiaquine; Zanzibar
MeSH Terms: conditions — Malaria, Falciparum | interventions — Artemether, Lumefantrine Drug Combination; Amodiaquine

STUDY DESIGN:
Intervention Model Description: A comparative randomised study comparing oral treatment with AQ + AS and CO of uncomplicated falciparum malaria in children.
Masking Description: The AQ+AS (AA) group received their drugs under direct observation once daily for 3 days. The Coartem (CO) group received their drugs twice daily, the second (evening) dose also under supervision. Drug treatment was thus not be blinded.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Artemether-lumefantrine (AL) (Active Comparator): One tablet of artemether-lumefantrine (Coartem®) was administered twice daily for 3 days to children with a body weight of 9 to <15 kg, and 2 tablets were administered twice daily for 3 days to children with a body weight of >15 to 25 kg. All doses were taken under direct observation.
  Interventions: Drug: Artemether-lumefantrine
- Artesunate + Amodiaquine (AA) (Active Comparator): Artesunate + amodiaquine (ASAQ) was administered as follows: 4 mg/kg body weight of artesunate plus 10 mg/kg body weight of amodiaquine once daily for 3 days under direct observation.
  Interventions: Drug: Coadministered Artesunate plus Amodiaquine

INTERVENTIONS:
Drug: Artemether-lumefantrine — Two doses a day for 3 days, under supervision
  Other Names: Coartem®
  Arms: Artemether-lumefantrine (AL)
Drug: Coadministered Artesunate plus Amodiaquine — One dose a day for 3 days, under supervision
  Arms: Artesunate + Amodiaquine (AA)

SUMMARY:
The primary objective of the study was to determine PCR corrected cure-rates up to day 42 in children with uncomplicated malaria, treated with either Artesunate + Amodiaquine or Coartem®.

Secondary objectives were to determine safety and possible selection of mutations related to the resistance of the tested drugs.

DETAILED DESCRIPTION:
Combination therapy, the new strategy for malaria treatment, is based on the hypothesis that two (or more) components of different mechanisms of action protect each other from development of resistance. Artemisinin as well as its two derivatives, e.g. artemether and artesunate, constitute a family of compounds with several attractive features for such a combination, due mainly to their rapid onset of effective action against multidrug-resistant P. falciparum and their gametocytocidal effect, which potentially reduces transmission of resistant alleles. There also appears to be no cross-resistance with other known anti-malarials. Because of the short half-life of this family of compounds, their use as mono-therapy requires multiple daily doses over a period of 7 days. Combining them with longer acting partner -drugs allows for a reduction in treatment duration while simultaneously enhancing the efficacy and reducing the likelihood of resistance development.

As of October 2001 the following anti-malarial drugs were recommended for malaria treatment in Zanzibar:

1. Artesunate (AS)+ Amodiaquine (AQ) - "first line" (AA)
2. Lumefantrine-artemether (Co-artem®) (CO) - "second line"
3. Quinine, if failure or contra indication of 1 & 2, or for treatment of severe malaria
4. Sulfadoxine-pyrimethamine (SP) for Intermittent Presumptive Treatment in pregnancy (IPT)

The move that the Zanzibar Ministry of Health has taken with this new treatment policy/strategy provided a unique opportunity to investigate the potential value of combination therapy when introduced on a large scale. Using artemisinine derivatives in combination with anti-malarials with longer half-lives is thought to be highly effective and considerably prevent the development of parasite resistance to the individual drugs. This study therefore provided baseline data on the efficacy of the new treatment policy and also for future monitoring of the policy in Zanzibar.

All children presenting with clinical signs of malaria at the study site were considered possible study subjects. The guardians of these children were informed about the study orally in Swahili for providing informed consent. Those who were willing to participate in the study were treated according to local standard procedure. The patient was tested for parasites using light microscopy on Giemsa stained blood films. A detailed clinical history, a clinical examination including an axillary temperature, was assessed. Haemoglobin was assessed and blood samples were collected on filter paper for each child for genotyping of the parasites as well as for determining blood levels of different antimalarial drugs.

The children included in the study were assigned to one of the two treatment options according to randomisation schedule, except children <9 months weighing <9 kg who were assigned AA because AL was registered for treatment of children <9 months weighing <9 kg. The drugs were given in standard doses according to bodyweight: artesunate 4 mg/kg bodyweight + amodiaquine 10 mg/kg bodyweight, once daily for 3 days, Coartem: 9 to <15 kg: 1 tablet; 15-25 kg: 2 tablets, twice daily for 3 days. All drugs were administrated under direct supervision of a study nurse. Full drug doses were re-administered if a patient spits out or vomits within 30 minutes. Drug treatment was provided free of charge.

The guardian was asked to bring their child back to the study site on day 1, 2, 3, 7, 14, 21, 28, 35 and 42. If they failed to do so they were visited in their homes to assure proper follow-up. At each follow-up the investigator asked about concomitant medication and adverse events, carefully filling out the clinical report form (CRF). If, during the follow-up between day 14 and 42, a child presented with fever, all tests and examinations were run as on day 0. If the child was clinically and parasitologically diagnosed with malaria again, he was treated as a new infection as of the national recommended guidelines. If diagnosed with severe malaria during the follow-up period the patient was given rescue treatment (oral or intravenous Quinine) and taken out of the study. Each time an enrolled child presented at the site the CRF was completed with regards to clinical and laboratory status, treatment given and possible adverse events.

The study drugs were obtained from the respective companies with the assistance of WHO/TDR and RBM.

ELIGIBILITY:
Inclusion Criteria:

* Children age 6-59 months and body weight ≥6 kg (AQ+AS); 9-59 months and body weight ≥9 kg (AL)
* Fever or history of fever in the preceding 24 hours
* Parasitemia ≥2000 ≤200.000 parasites per µl
* Informed consent given by the child's parent or other adult guardian

Exclusion Criteria:

* Signs of severe malaria or other danger signs, such as: 1.Unconsciousness; 2. Not able to sit or stand; 3.Severe anaemia (Hb ≤ 5 g/dl); 4.Convulsions; 5. Shock (systolic BP<50 mmHg); 6. Not able to drink or breastfeed; 7. Vomiting 3 times or more the past 24 hrs
* Other diseases associated with fever
* History of allergy to test drugs
* History of intake of any drugs other than paracetamol and aspirin within 3 days

Ages: 6 Months to 59 Months | Sex: All
Age Groups: Child
Enrollment: 408 (Actual)
Dates: Start 2002-11-01 (Actual); Primary Completion 2003-02-17 (Actual); Study Completion 2003-02-17 (Actual)

PRIMARY OUTCOMES:
PCR corrected cure-rates up to day 42 in children with uncomplicated malaria, treated with either Artesunate + Amodiaquine (AA) or Coartem® (CO) | 42 days
  Comparing PCR adjusted parasitological cure rate (PCR-APCR) between the two treatment options up to day 42. Parasitological cure will be adjusted using PCR genotyping of msp2 marker. Recrudescence is defined as the presence of at least one matching allelic band, and reinfection as the absence of any matching allelic band on day 0 and day of recurring parasitaemia. Patients with recurrent parasitaemia having missing filter paper sample or negative PCR results will be considered uncertain with regards to PCR adjusted outcome.

SECONDARY OUTCOMES:
Safety of treatment with Artesunate + Amodiaquine (AA) or Coartem® (CO): Proportion of subjects with adverse events | 42 days
  Proportion of subjects with adverse events, including early vomiting and mean values of white blood cells (WBC) and neutrophils
Parasite clearance | 42 days
  Proportion of patients with microscopy detectable parasitaemia at each time point
Gametocyte carriage | 42 days
  Proportion of patients with microscopy detectable gametocytes at each time point
Fever clearance | 42 days
  Proportion of patients with fever at each time point
Hemoglobin | 42 days
  Mean and individual hemoglobin values at different time points during follow up
Selection of mutations in P. falciparum related to the resistance of the study drugs | 42 days
  Change in possible selections of mutations related to quinoline resistance. Percentage of pfcrt and pfmdr1 mutations on day 0 and day of recurrent infection.

CONTACTS AND LOCATIONS:
Overall Officials: Abdullah Ali, Principal Investigator — Zanzibar Malaria Control Programme

REFERENCES:
- [Result] Martensson A, Stromberg J, Sisowath C, Msellem MI, Gil JP, Montgomery SM, Olliaro P, Ali AS, Bjorkman A. Efficacy of artesunate plus amodiaquine versus that of artemether-lumefantrine for the treatment of uncomplicated childhood Plasmodium falciparum malaria in Zanzibar, Tanzania. Clin Infect Dis. 2005 Oct 15;41(8):1079-86. doi: 10.1086/444460. Epub 2005 Sep 13. PMID 16163624
- [Result] Sisowath C, Ferreira PE, Bustamante LY, Dahlstrom S, Martensson A, Bjorkman A, Krishna S, Gil JP. The role of pfmdr1 in Plasmodium falciparum tolerance to artemether-lumefantrine in Africa. Trop Med Int Health. 2007 Jun;12(6):736-42. doi: 10.1111/j.1365-3156.2007.01843.x. PMID 17550470
- [Result] Holmgren G, Hamrin J, Svard J, Martensson A, Gil JP, Bjorkman A. Selection of pfmdr1 mutations after amodiaquine monotherapy and amodiaquine plus artemisinin combination therapy in East Africa. Infect Genet Evol. 2007 Sep;7(5):562-9. doi: 10.1016/j.meegid.2007.03.005. Epub 2007 Mar 31. PMID 17467344